CLINICAL TRIAL: NCT00615160
Title: Phase II Randomized, Parallel-Group Trial on PTK-ZK With or Without DTIC in Patients With Non-resectable Metastatic Malignant Melanoma
Brief Title: PTK/ZK in Disseminated Malignant Melanoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Substance was withdrawn from further development.
Sponsor: Michael Weichenthal (Other)
Responsible Party: Sponsor-Investigator, Michael Weichenthal, Senior Consultant, University Hospital Schleswig-Holstein
Organization: University Hospital Schleswig-Holstein (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UKSH A-105; EudraCT No. 2005-002192-32
Record Dates: First submitted 2008-01-31; First posted 2008-02-14 (Estimated); Last update posted 2021-10-06 (Actual); Status verified 2021-09

CONDITIONS: Melanoma
Keywords: Metastatic melanoma; anti angiogenetic treatment
MeSH Terms: conditions — Melanoma | interventions — vatalanib; Dacarbazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): PTK787/ZK 222584 (PTK-ZK) taken orally with a daily flat dose of 1250 mg on days 1 to 28 (= 1 cycle)
  Interventions: Drug: PTK787/ZK 222584
- B (Experimental): combined treatment with DTIC 850 mg/m² on day 1 + PTK-ZK 1250 mg flat dose on days 1 to 28
  Interventions: Drug: PTK787/ZK 222584; Drug: Dacarbazine

INTERVENTIONS:
Drug: PTK787/ZK 222584 — PTK-ZK capsules taken orally with a daily flat dose of 1250 mg
Drug: Dacarbazine — Dacarbazine 850 mg/m² on day 1 q4w
  Other Names: DTIC
  Arms: B

SUMMARY:
To evaluate the efficacy of PTK-ZK on metastatic melanoma either as a single agent treatment or in combination with standard chemotherapy according to RECIST criteria. Further to evaluate the safety and tolerability of PTK-ZK in patients with metastatic melanoma either as a single agent treatment or in combination with standard chemotherapy

DETAILED DESCRIPTION:
This is a multicenter, randomized, open-label, parallel-group phase II study to evaluate the efficacy and safety of PTK-ZK in the treatment of patients with metastatic malignant melanoma who do not qualify for surgical resection:

* progressive locoregionary disease not to be controlled by surgical measures
* distant metastasis other than brain metastasis not eligible for surgical resection or radiotherapy All patients will be treated with PTK-ZK 1250mg administered orally once a day for treatment cycles of 28 days. In case of unacceptable toxicity the dose can be reduced to 1000 mg and further on to 750 mg daily.

Patients in Arm B additionally receive intravenous DTIC 850mg/m² on day 1 of each cycle.

After informed consent is given by the patient a biopsy from a metastasis should be taken before the first intake of study medication and at the end of cycle 2 to specify markers of angiogenesis and MVD (Micro vessel density).

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed nonresectable metastatic melanoma Stage III or IV (AJCC 2002) including patients with unknown primary melanoma,
* Progressive disease, defined as an increase of tumour volume according to RECIST criteria, within the last 6 months,
* Fulfilling the minimum RECIST requirements for evaluation of tumor response,
* At least two cutaneous or soft tissue lesions that can be biopsised prior to and after treatment, respectively,
* Able to undergo either contrast-enhanced CT scan or contrast-enhanced MRI scan for tumor assessment,
* Life expectancy greater than 3 months,
* ECOG performance status <2,
* Age > 18 years,
* Able to swallow and retain intact investigational drug tablets,
* Willingness and ability to adhere to the study requirements as outlined in the protocol,
* Agreement to use a highly effective method of birth control throughout the study period and 3 months thereafter for sexually active males and females of childbearing potential. Barrier contraceptives must be used throughout the trial. Oral, implantable, or injectable contraceptives may be affected by cytochrome P450 interactions, and are therefore not considered effective for this study.
* Able to provide informed consent.

Exclusion Criteria:

* One or more previous systemic therapies for metastatic melanoma, excluding prior systemic therapy given for high-risk primary tumor, lymph node metastasis, or other regional (AJCC stage III) disease spread as postoperative adjuvant therapy.
* Anticancer therapy (chemotherapy, radiotherapy, vaccines, immunotherapy, and hormone therapy) delivered within 4 weeks prior to the 1st dose of study drug, and 2 weeks prior for palliative "spot" radiotherapy to bone metastases),
* History of uveal melanoma,
* Female patients who are pregnant or breast feeding. Women of childbearing potential must have a negative serum pregnancy test 48 hours prior to administration of study treatment.
* Impaired organ and bone marrow function defined as one or more of the following:
* Absolute neutrophil count (ANC) <1,500/µl,
* Platelets <100,000/µl,
* Total bilirubin >1.5 x ULN,
* ASAT (SGOT)/ALAT (SGPT) > 3x ULN (5x if liver metastases are present)
* History or presence of central nervous system (CNS) disease (i.e., primary brain tumor, malignant seizures, CNS metastases or carcinomatous meningitis)
* Another malignancy in the 5 years prior to enrollment other than non melanoma skin cancer, or cervix carcinoma in situ,
* Major Surgery < 10 days prior to the start of study treatment
* Inadequate recovery from previous surgery, radiation, chemo-, biologic or immunotherapy
* Ongoing effects from previous investigational drug studies or concomitant participation in other investigational drug studies
* Prior use of PTK-ZK or other VGEF receptor antagonists,
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to PTK-ZK, or patients who have known hypersensitivity to the study medication
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of PTK/ZK (i.e., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, bowel obstruction, or inability to swallow the tablets).
* Myocardial infarction ≤ 6 months prior to randomization
* Acute or chronic liver disease (i.e., hepatitis, cirrhosis)
* Uncontrolled high blood pressure, history of labile hypertension, or history of poor compliance with an antihypertensive regimen
* Chronic renal disease, i.e. Creatinine >1.5 x upper limit of normal (ULN) OR Proteinuria based on dip stick reading positive > +1 OR if the dip stick result is +1, total urinary protein > 500 mg and measured creatinine clearance < 50 ml/min from a 24-hour urine collection Haemoglobin < 9 g/dL (patients may be transfused to achieve Hb > 9 g/dL)

Other uncontrolled concomitant condition, including but not limited to:

* ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, serious uncontrolled cardiac arrhythmia, uncontrolled diabetes, seizure disorder
* Psychiatric illness/social situations that would limit compliance with study requirements, or other conditions that compromise the patient's ability to understand the patient information, to give informed consent, to comply with the trial protocol, or to complete the study
* Human immunodeficiency virus (HIV) infection,
* Prior enrollment into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2006-12; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Overall response defined by RECIST criteria | 8 week response rate

SECONDARY OUTCOMES:
Toxicity and safety | continuously
Tumor control as defined by the number of patients with objective tumor response or tumor stabilization according to RECIST criteria | Best response during time of treatment
Time to progression | Time of progression
Quality of life (EORTC QLQ C30) | During active treatment

CONTACTS AND LOCATIONS:
Overall Officials: Michael Weichenthal, MD, Study Director — UK-SH Department of Dermatology
Locations (4):
- Germany (4):
  - Dpt. of Dermatology, University of Cologne, Cologne
  - Dpt. of Dermatology, University of Essen, Essen
  - Dpt. of Dermatology, University of Frankfurt, Frankfurt am Main
  - Dpt. of Dermatology; UK-SH Campus Kiel, Germany, Kiel